CLINICAL TRIAL: NCT00003267
Title: A Randomized Phase III Trial for Evaluation of Usefulness of Pelvic Drains After Radical Hysterectomy and Node Dissection (RHND)
Brief Title: Pelvic Drains After Radical Hysterectomy in Treating Patients With Uterine, Cervical, or Vaginal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: EORTC-55962; EORTC-55962
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Cervical Cancer; Endometrial Cancer; Infection; Perioperative/Postoperative Complications; Vaginal Cancer
Keywords: stage I cervical cancer; stage II cervical cancer; stage I vaginal cancer; stage II vaginal cancer; stage I endometrial carcinoma; stage II endometrial carcinoma; infection; perioperative/postoperative complications
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Infections; Postoperative Complications; Vaginal Neoplasms | interventions — Therapeutics; Surgical Procedures, Operative

INTERVENTIONS:
Procedure: infection prophylaxis and management
Procedure: management of therapy complications
Procedure: surgical procedure

SUMMARY:
RATIONALE: The use of pelvic drains may help to prevent complications following radical hysterectomy and pelvic lymphadenectomy. It is not known whether receiving pelvic drains during surgery is more effective than receiving no pelvic drains during surgery in patients with uterine, cervical, or vaginal cancer.

PURPOSE: Randomized phase III trial to determine if the use of pelvic drains following radical hysterectomy and pelvic lymphadenectomy is effective in treating patients with uterine, cervical, or vaginal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate postoperative complications associated with the use or omission of pelvic drains following radical hysterectomy and node dissection that includes suturing of the vaginal cuff and no peritonealization.

OUTLINE: This is a randomized, two-arm study. All patients receive radical hysterectomy (Rutledge-Piver II-III type) and pelvic lymphadenectomy, without pelvic and parietal peritonealization, with suturing of the vaginal cuff and closure of fascia and cutaneous layers; lumboaortic node dissection is optional. Patients are randomized during surgery to one of two arms: those on arm I receive pelvic drains and those on arm II do not. Those in arm I have drains applied in the pelvis, and lymph is collected by vaginal and/or transabdominal drains located in both retroperitoneal fossa. Drains are removed when the loss is less than 50 mL in 24 hours. Patients in both arms are followed at 2-3 months and 12 months after surgery.

PROJECTED ACCRUAL: 214 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven cervical, vaginal, or endometrial carcinoma for which abdominal radical hysterectomy (Rutledge-Piver II or III type) and pelvic node dissection is indicated The following are excluded: Extensive intraoperative retroperitoneal blood loss (more than 3000 mL) Excessive postsurgical hemorrhage or oozing of the wound area requiring postoperative drainage Concurrent urinary or bowel injury/deviation or surgical procedures for urinary incontinence (Burch etc.) Application of prophylactic abdominal mesh for subsequent radiotherapy

PATIENT CHARACTERISTICS: Age: Not specified Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior neoadjuvant chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 1998-02; Primary Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio L. Pecorelli, MD, Study Chair — Spedali Civili di Brescia
Locations (18):
- Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Institut Gustave Roussy, Villejuif, France
- University Medical Center, Freiburg im Breisgau, Germany
- Italy (7):
  - Universita di Brescia, Brescia
  - Instituto Scientifico H.S. Raffaele, Milano (Milan)
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan)
  - Azienda Ospedaliera Di Parma, Parma
  - University and I.R.C.C.S. Policlinico San Matteo, Pavia
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Civile, Voghera (PV)
- Netherlands (4):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Utrecht, Utrecht
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Instituto Valenciano De Oncologia, Valencia, Spain

REFERENCES:
- [Result] Franchi M, Trimbos JB, Zanaboni F, v d Velden J, Reed N, Coens C, Teodorovic I, Vergote I. Randomised trial of drains versus no drains following radical hysterectomy and pelvic lymph node dissection: a European Organisation for Research and Treatment of Cancer-Gynaecological Cancer Group (EORTC-GCG) study in 234 patients. Eur J Cancer. 2007 May;43(8):1265-8. doi: 10.1016/j.ejca.2007.03.011. Epub 2007 Apr 26. PMID 17466514